CLINICAL TRIAL: NCT01874613
Title: Clinical Study of Skull Defect Reconstruction With Patient-specific Fibre-reinforced Composite Implant
Brief Title: Clinical Study of FRC Implant to Treat Skull Bone Defects
Acronym: Cranio-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: Oulu University Hospital (Other); Turku Clinical Biomaterials Centre (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T97/2011
Record Dates: First submitted 2012-11-13; First posted 2013-06-11 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Cranial Bone Defect; Orbital Base Fracture
Keywords: Craniofacial bone reconstruction; Fibre-reinforced composite; Bioactive glass; Craniotomy; Skull bone defect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Skull bone reconstruction (Experimental): Patients with skull bone defect
  Interventions: Device: FRC implant reconstruction
- Orbital floor defect (Experimental): Patients with orbital floor defect
  Interventions: Device: FRC implant reconstruction

INTERVENTIONS:
Device: FRC implant reconstruction — A cranioplasty with the FRC implant is performed.
  Arms: Skull bone reconstruction
Device: FRC implant reconstruction — The orbital floor fracture is reconstructed with the FRC implant.
  Arms: Orbital floor defect

SUMMARY:
Bioactive fibre-reinforced composite implant is used for reconstruction of skull bone defects and orbital floor defects.

Functional and aesthetic outcome is assessed by patient and doctor.

DETAILED DESCRIPTION:
Development phase: Clinical trial Objectives: Assessment of functional and aesthetic outcome Methodology: Intervention study Sample size: 35+20+25 Main criteria for inclusion: Skull bone defect OR orbital floor fracture

Investigational drug/treatment, dose and mode of administration: FRC implant Comparative drug(s)/placebo/treatment, dose and mode of administration: -

Duration of treatment: 2 years of follow-up

Assessments:

Clinical outcome and radiologic assesment Functional and aesthetic outcome with Visual Analog Scale (VAS). Pain assessment with VAS.

Statistical methods:

Adequate statistical methods for publishing in international peer-reviewed journals.

ELIGIBILITY:
Inclusion Criteria:

Study arm 1:

* patients with skull bone defect
* reconstruction indications fullfilled

Study arm 2:

* patients with orbital floor defect
* reconstruction indication fullfilled

Exclusion Criteria:

* if informed consent cannot be obtained

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-01; Primary Completion 2016-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Functional outcome (a composition of following measures) | 2 year follow-up
  After reconstruction, patient follow-up protocol follows to assess functional outcome, including safety.
  Follow-up is done at timepoints of 1 week, 1 month, 3 months, 6 months and after that every 6 month up to 2 years post-operatively. After this the follow-up is continued yearly, if necessary.
  Visual and manual assessment is done by a doctor. Lateral and PA skull rtg is obtained to assess the fixation and position of the implant.
  C-reactive protein level and leukocyte level is measured to assess the possible inflammation.

SECONDARY OUTCOMES:
Aesthetic outcome (a composition of following measures) | 2 years post-operatively
  After reconstruction, patient follow-up protocol follows to assess aesthetic outcome.
  Follow-up is done at timepoints of 1 week, 1 month, 3 months, 6 months and after that every 6 month up to 2 years post-operatively. After this the follow-up is continued yearly, if necessary.
  Visual and manual assessment is done by a doctor. Visual Analog Scale (VAS) is used by patient to assess
  * functional outcome
  * aesthetic outcome
  * pain Lateral and PA skull rtg is obtained to assess the fixation and position of the implant.
  C-reactive protein level and leukocyte level is measured to assess the possible inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Kalle J Aitasalo, Professor, Principal Investigator — Turku University Hospital
Locations (1):
- Department of Otorhinolaryngology, Turku, N/A = Not Applicable, Finland